CLINICAL TRIAL: NCT00270842
Title: Effect of Exercise on Gait and Balance in Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: O4006-R
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Results first posted 2015-04-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Diabetic Neuropathies; Peripheral Nerve Diseases; Peripheral Nervous System Diseases
Keywords: Education; Exercise; Gait; Peripheral Nervous System; Postural Balance; Self Efficacy; Tai Chi Chuan
MeSH Terms: conditions — Diabetic Neuropathies; Peripheral Nervous System Diseases; Motor Activity | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Education Control Group (Placebo Comparator): Education group that is the control group for the study. Is a 10 week course with diverse health education topics.
  Interventions: Behavioral: Education Control group
- Functional Balance Training (Experimental): Exercise group that participated in functional balance training
  Interventions: Behavioral: Functional Balance
- Tai chi (Experimental): Exercise Group that participated in tai chi training classes
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Tai Chi — This intervention is a 10 week Tai Chi group exercise class designed specifically for persons with Peripheral Neuropathy, having difficulty feeling their feet.
  Arms: Tai chi
Behavioral: Functional Balance — This intervention is a 10 week Functional Balance group exercise class designed specifically for persons with Peripheral Neuropathy, having difficulty feeling their feet.
  Arms: Functional Balance Training
Behavioral: Education Control group — This control group participated in 10 weeks of general health education classes.
  Arms: Education Control Group

SUMMARY:
The purpose of this study is to find out if participation in one of the study groups: functional balance training, Tai Chi, or education, results in better outcomes overall. The outcomes that we are primarily interested in are related to walking ability and balance.

DETAILED DESCRIPTION:
Since the 1970's, researchers and epidemiologists have documented that patient falls are a high-risk, high volume, high cost adverse events contributing to morbidity, mortality, decreased quality of life, and premature nursing home placement. Despite thousands of research studies published on patient falls, few studies have focused on the effectiveness of interventions , and fall rates and associated injuries among the elderly continue to rise. Impaired gait and balance (referred to as impaired stability) is one of the most significant causes and consequences of falls. Persons with peripheral neuropathy represent one of the largest patient populations with impaired stability. Lower limb peripheral neuropathy (LLPN) includes sensory and motor impairments that result in impaired gait and balance, jeopardizing safe mobility. Emerging evidence suggests that exercise programs can be effective in improving gait and balance in general fall risk populations, as well as reducing falls and fall-related injuries. Exercise interventions have been designed to reduce fall risk and promote successful aging. These interventions come in many forms, but the most common interventions are exercise training and Tai Chi, offered individually and in small group formats. Further research is needed to gain insight into the underlying mechanisms of different type of exercises and their impact on stability in veterans with LLPN. Research is needed to determine the type or combination of types of exercise to produce a more normal and/or stable gait in this high-risk patient population. Researchers are beginning to document that exercise interventions positively influence a person's fall self efficacy, i.e. self confidence for avoiding a fall, an important factor in understanding and examining a persons' behaviors related to fall risks. The emphasis on functionally based interventions has led to inappropriate broad groupings of older persons with mobility disorders. A weakness of previous studies was that they aggregated heterogeneous patient populations, resulting in neurological and musculoskeletal diagnostic heterogeneity and the confounding of results. Focusing on a homogeneous patient population is necessary to distinguish unique sensory, gait and balance deficits that contribute to impaired stability and mobility risk, as well as to better understand unique responses to treatment that are clouded when diverse patients are aggregated. We will target veterans with LLPN--one of the largest groups of patients referred to our Falls Clinic, and an understudied population with respect to safe patient mobility. This will allow us to design targeted interventions likely to be more effective than those tested on heterogeneous elderly populations, where visual and vestibular input to compensate for impaired proprioception were not taken into account.

The goal of this study is to improve successful adaptation to aging and quality of life in veterans with lower limb peripheral neuropathy (LLPN). Functional Balance Training and Tai Chi, the two exercise interventions tested in this study, have been documented to improve gait and balance, and decrease falls and associated fall-related injuries in the general elderly population. We are interested in whether one or both of these exercise interventions (successful in general elderly populations) would be effective in a special subpopulation of elderly, namely persons with LLPN.

The purpose of this study is to compare the effectiveness of these two exercise interventions and an education control group. Effectiveness will be assessed by studying the impact of interventions on (1) composite measures of stability (gait and balance), (2) fall self-efficacy, and (3) patient acceptance. Given the well-documented links between falls and fall-related injuries (ultimate outcomes) our study will focus on stability (intermediate outcome). Because falls and fall-related injuries are relatively rare events, examining stability as an outcome will allow us to have sufficient power to test our hypotheses with a relatively small sample size thereby decreasing the cost and duration of the study without sacrificing the rigor of the research design.

ELIGIBILITY:
Inclusion Criteria:

* Corrected vision not worse than 20/50 to have visual acuity to read and follow instructions.
* Ability to ambulate household distances with or without an assistive device. This reflects a minimum functional status for ambulation as primary mode of mobility.
* Symptoms and Signs consistent with LLPN as determined by the Michigan Diabetic Neuropathy Scale (Score greater than 6, presence of mild PN). The Michigan Diabetic Neuropathy Score quantifies sensory impairment, muscle strength, and reflexes, using vibration, filament, pin prick, and physical touch. Scale ranges from 0-46, with higher score indicating great severity of PN. The score is used to stratify severity of PN, and takes approximately 10-15 minutes to complete. Testing aspects elicit sensation from small and moderate nerve fibers, and is more sensitive to mild to moderate sensory neuropathy. This test was selected rather than the gold standard EMG in order to screen for study subjects, is less invasive, and reduces the burden of subject screening for inclusion into this study.

Exclusion Criteria:

* Cognitive impairment with MMSE score less than 24, level 24 and below scores indicated cognitive impairments, limiting ability to remember instructions.
* Metastatic cancer, limits ability to complete the intensity and duration of the study.
* Central neurological dysfunction e.g. diagnosis of hemiparesis, cerebellar dysfunction, Parkinson's disease as determined by medical record review. These neurological impairments impair gait and balance, and would jeopardize safety if randomized to an intervention group.
* Lower extremity amputation, a physical disability that results in altered postural balance.
* Lower extremity abnormality other than peripheral neuropathy, such as foot drop, as participation in class would compromise patient safety.
* Mobility limitations due to altered lower extremity skin integrity/ulcer, where pain would limit gait and weight-bearing would be contraindicated such as stasis and foot ulcers or claudication.
* Medically unstable upon exam, i.e. poorly controlled blood pressure and blood sugar, coronary artery disease, where group participation would compromise medical status.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Quigley, PhD MPH, Principal Investigator — James A. Haley Veterans Hospital
Locations (1):
- James A. Haley Veterans Hospital, Tampa, Florida, United States

REFERENCES:
- [Result] Quigley PA, Bulat T, Schulz B, Friedman Y, Hart-Hughes S, Richardson JK, Barnett S. Exercise interventions, gait, and balance in older subjects with distal symmetric polyneuropathy: a three-group randomized clinical trial. Am J Phys Med Rehabil. 2014 Jan;93(1):1-12; quiz 13-6. doi: 10.1097/PHM.0000000000000052. PMID 24355993

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Education Control Group | Functional Balance Training | Tai Chi
Started | 33 | 34 | 34
Completed | 18 | 18 | 18
Not Completed | 15 | 16 | 16

BASELINE CHARACTERISTICS:
Population: 101 subjects were enrolled, however, 2 subjects dropped after completion of baseline assessments. Only 99 are included in the data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Education Control Group | Functional Balance Training | Tai Chi | Total
Number analyzed (Participants) | 31 | 34 | 34 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (10.2) | 67.6 (10.6) | 68.4 (9.3) | 67.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 5 | 15
  Male | 25 | 30 | 29 | 84

OUTCOME MEASURES:

1. Primary Outcome: Gait and Balance Measures
Description: The Berg Balance Scale is a commonly used clinical, performance-based measure designed to evaluate performance during various balance activities in community dwelling and institutionalized older adults. The scale consists of 14 common daily balance tasks. Administration requires only minimal basic equipment and takes approximately 15 minutes. All 14 sub-tests are scored on a 5-point ordinal scale based on the subject's ability to perform the requested task safely and in a timely manner. Sub-test scores are summed to achieve a total score ranging from 0 to 56 with higher scores indicating better performance.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Control Group | Functional Balance Training | Tai Chi
Number analyzed (Participants) | 31 | 34 | 34
units on a scale | 51.3 (5.4) | 51.2 (7.0) | 52.3 (3.3)

2. Secondary Outcome: Fall Self Efficacy
Description: Fall Self Efficacy is operationalized as perceived self efficacy (i.e. self confidence) for avoiding a fall during 10 global, relatively non-hazardous activities of daily living (getting dressed and undressed, for example). Fall self efficacy manifests itself with different degrees of fear of falling, each with a unique associated risk level. The MFES is simple, quick, easy-to-administer scale that assesses a patient's self-reported ability to perform, without falling, each of 14 common activities of daily living in a Likert scale format. Total scale ranges from 0 to 140, the higher score indicated more confidence in ability to manage a fall.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Control Group | Functional Balance Training | Tai Chi
Number analyzed (Participants) | 33 | 34 | 34
units on a scale | 121.5 (19.9) | 113.7 (32.3) | 123.1 (27.3)

ADVERSE EVENTS:
Time Frame: From enrollment to end of study participation.
Arm/Group | Education Control Group | Functional Balance Training | Tai Chi
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/31 | 0/34 | 0/34

LIMITATIONS AND CAVEATS:
Due to the large number of drop outs following the 10 week data point, maintenance of gait and balance changes is uncertain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No